CLINICAL TRIAL: NCT04107129
Title: Predicting Endometrial Receptivity for Optimal Reproductive Management (PERFORM)
Brief Title: Predicting Endometrial Receptivity for Optimal Reproductive Management
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Professor, Obstetrics and Gynecology, Stanford University
Other Study IDs: 51702; 4R44HD097750-02 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-07

CONDITIONS: Infertility, Female; Endometriosis
Keywords: Infertility; Endometriosis; BLC6; SIRT1; In Vitro Fertilization (IVF); Embryo Transfer (ET); Frozen Embryo Transfer (FET); Assisted Reproductive Technology (ART); PERFORM
MeSH Terms: conditions — Infertility, Female; Endometriosis; Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometrial biopsy will be collected. Urine, saliva, and blood samples will also be collected for future studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Known Endometriosis: Known Endometriosis undergoing IVF with PGTA
  Interventions: Procedure: Endometrial Biopsy; Other: Euploid embryo transfer; Diagnostic Test: Blood sample
- Unexplained Infertility: Unexplained Infertility undergoing IVF with PGTA
  Interventions: Procedure: Endometrial Biopsy; Other: Euploid embryo transfer; Diagnostic Test: Blood sample
- Low Risk Controls: Low Risk Controls undergoing IVF with PGTA
  Interventions: Procedure: Endometrial Biopsy; Other: Euploid embryo transfer; Diagnostic Test: Blood sample

INTERVENTIONS:
Procedure: Endometrial Biopsy — An endometrial biopsy is the removal of a small piece of tissue from the endometrium, which is the lining of the uterus. Endometrial tissue will be tested for BCL6 and SIRT1 Biomarkers
Other: Euploid embryo transfer — Patients undergoing IVF and Preimplantation genetic testing will undergo delayed euploid frozen embryo transfer per clinical protocol and standard of care.
Diagnostic Test: Blood sample — Estradiol and Progesterone levels in the blood will be checked

SUMMARY:
The purpose of this study is to understand why some women are infertile (unable to conceive a child). The investigators hope to learn if an endometrial biopsy after egg retrieval is feasible for detecting biomarkers for endometriosis and predicting implantation and pregnancy rate after embryo transfer.

This study design will provide for the first time, an opportunity to compare endometrial biopsy material from hyperstimulated (gonadotropin treated) subjects after egg retrieval. If successful, it would provide a new protocol for women with unexplained infertility or those with known endometriosis to avoid poor IVF outcomes.

DETAILED DESCRIPTION:
The investigators will recruit 100 women who are undergoing IVF with egg retrieval and delayed embryo transfer to consent to endometrial biopsy 1 week after egg retrieval. Currently most women in the Stanford's IVF program undergo egg retrieval with delayed embryo transfer (ET) with preimplantation genetic testing of embryos. This delay allows most to avoid the condition known as ovarian hyperstimulation and allows time for genetic screening (PGT-A) performed on embryos. Such a delay also opens the window for endometrial assessment for proteins like SIRT1 and BCL6 that have been suggested to be associated with endometriosis. Endometriosis is thought to cause IVF failure (Littman et al., 2002); by treating endometriosis in the future, clinicians might avoid IVF failure due to an unexpected non-receptive endometrium (Littman et al., 2002). This study design will provide for the first time, an opportunity to compare endometrial biopsy material from hyperstimulated (gonadotropin treated) subjects after egg retrieval. If successful, it would provide a new protocol for women with unexplained infertility or those with known endometriosis to avoid poor IVF outcomes.

There is some evidence that endometrial scratching (biopsy) may enhance embryo attachment in future cycles (Vitagliano et al., 2018), although not all studies agree (Lensen et al., 2019). The endometrial biopsy taken in the secretory phase will be tested for BCL6 and SIRT1 expression, two proteins highly associated with the presence of endometriosis (Yoo et al., 2017). The samples of endometrium will be processed (put into formalin and paraffin blocks or saved in RNA later and not be analyzed until after completion of the ART cycle. Patients as well as the clinicians will be blinded to results and until the conclusion of the ART cycle following embryo transfer and subsequent pregnancy testing. This will be done to avoid interfering with the current ART cycle and to avoid the introduction of bias. Patients will be provided with test results after completion of the first embryo transfer if they wish to know.

ELIGIBILITY:
Inclusion Criteria:

1. Age - 18 to 42
2. AMH ≥ 1
3. Planning to undergo IVF with delayed embryo transfer
4. Must have blastocyst(s) by day 6 that were biopsied for PGT-A
5. BMI 18-35

Exclusion Criteria:

1. Uterine fibroids > 4 cm in size
2. Polycystic ovary syndrome (PCOS) according with the Rotterdam criteria.
3. Ovarian failure and subjects receiving donor oocytes/embryos
4. Anti-cardiolipid and/or lupus anti-coagulant abnormalities by history
5. Diabetes mellitus (Type I or Type II)
6. Untreated hypothyroidism
7. Hyperprolactinemia
8. Uncorrected uterine anomaly

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult females of reproductive age.
Study Population: These criteria are meant to define two populations of women (high and low risk for endometriosis) and not include confounding diagnoses including PCOS, autoimmune conditions and endocrine disorders such as hypothyroidism and hyperprolactinemia.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
SIRT1 gene expression in the endometrium | 2-3 years
  Endometrial biopsy specimens will be stained for SIRT1 using immunostaining and Hscore assignment.

SECONDARY OUTCOMES:
BCL6 expression in the endometrium | 2-3 years
  Endometrial biopsy specimens will be stained for BCL6 using immunostaining and Hscore assignment.
Number of patients who have a positive pregnancy test (HCG level > 5) 9 days after embryo transfer | 2-3 years
  pregnancy rate
Number of embryo transfers that lead to live births | 2-3 years
  live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Ruth B Lathi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Fertility and Reproductive Health, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No
No PHI will be shared with collaborators. Collaborators will only have access to aggregate data by study group

REFERENCES:
- [Background] Budwit-Novotny DA, McCarty KS, Cox EB, Soper JT, Mutch DG, Creasman WT, Flowers JL, McCarty KS Jr. Immunohistochemical analyses of estrogen receptor in endometrial adenocarcinoma using a monoclonal antibody. Cancer Res. 1986 Oct;46(10):5419-25. PMID 3756890
- [Background] Simoens S, Dunselman G, Dirksen C, Hummelshoj L, Bokor A, Brandes I, Brodszky V, Canis M, Colombo GL, DeLeire T, Falcone T, Graham B, Halis G, Horne A, Kanj O, Kjer JJ, Kristensen J, Lebovic D, Mueller M, Vigano P, Wullschleger M, D'Hooghe T. The burden of endometriosis: costs and quality of life of women with endometriosis and treated in referral centres. Hum Reprod. 2012 May;27(5):1292-9. doi: 10.1093/humrep/des073. Epub 2012 Mar 14. PMID 22422778
- [Background] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Background] Endometriosis exerts "profound" economic burden in the US. (2007). PharmacoEconomics & Outcomes News. https://doi.org/10.2165/00151234-200705230-00025
- [Background] Evans-Hoeker E, Lessey BA, Jeong JW, Savaris RF, Palomino WA, Yuan L, Schammel DP, Young SL. Endometrial BCL6 Overexpression in Eutopic Endometrium of Women With Endometriosis. Reprod Sci. 2016 Sep;23(9):1234-41. doi: 10.1177/1933719116649711. Epub 2016 May 24. PMID 27222232
- [Background] Fox C, Morin S, Jeong JW, Scott RT Jr, Lessey BA. Local and systemic factors and implantation: what is the evidence? Fertil Steril. 2016 Apr;105(4):873-84. doi: 10.1016/j.fertnstert.2016.02.018. Epub 2016 Mar 3. PMID 26945096
- [Background] Lensen S, Osavlyuk D, Armstrong S, Stadelmann C, Hennes A, Napier E, Wilkinson J, Sadler L, Gupta D, Strandell A, Bergh C, Vigneswaran K, Teh WT, Hamoda H, Webber L, Wakeman SA, Searle L, Bhide P, McDowell S, Peeraer K, Khalaf Y, Farquhar C. A Randomized Trial of Endometrial Scratching before In Vitro Fertilization. N Engl J Med. 2019 Jan 24;380(4):325-334. doi: 10.1056/NEJMoa1808737. PMID 30673547
- [Background] Lessey BA, Metzger DA, Haney AF, McCarty KS Jr. Immunohistochemical analysis of estrogen and progesterone receptors in endometriosis: comparison with normal endometrium during the menstrual cycle and the effect of medical therapy. Fertil Steril. 1989 Mar;51(3):409-15. doi: 10.1016/s0015-0282(16)60545-9. PMID 2646155
- [Background] Lessey BA, Palomino WA, Apparao KB, Young SL, Lininger RA. Estrogen receptor-alpha (ER-alpha) and defects in uterine receptivity in women. Reprod Biol Endocrinol. 2006;4 Suppl 1(Suppl 1):S9. doi: 10.1186/1477-7827-4-S1-S9. PMID 17118173
- [Background] Likes CE, Cooper LJ, Efird J, Forstein DA, Miller PB, Savaris R, Lessey BA. Medical or surgical treatment before embryo transfer improves outcomes in women with abnormal endometrial BCL6 expression. J Assist Reprod Genet. 2019 Mar;36(3):483-490. doi: 10.1007/s10815-018-1388-x. Epub 2019 Jan 4. PMID 30610661
- [Background] Littman E, Giudice L, Lathi R, Berker B, Milki A, Nezhat C. Role of laparoscopic treatment of endometriosis in patients with failed in vitro fertilization cycles. Fertil Steril. 2005 Dec;84(6):1574-8. doi: 10.1016/j.fertnstert.2005.02.059. PMID 16359945
- [Background] Meyer WR, Lessey BA, Castelbaum AJ. Hydrosalpinx and altered uterine receptivity. Fertil Steril. 1997 Nov;68(5):944-5. doi: 10.1016/s0015-0282(97)90360-5. No abstract available. PMID 9389833
- [Background] Newcombe RG. Two-sided confidence intervals for the single proportion: comparison of seven methods. Stat Med. 1998 Apr 30;17(8):857-72. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-e. PMID 9595616
- [Background] Revised American Society for Reproductive Medicine classification of endometriosis: 1996. Fertil Steril. 1997 May;67(5):817-21. doi: 10.1016/s0015-0282(97)81391-x. No abstract available. PMID 9130884
- [Background] Schmittgen TD, Livak KJ. Analyzing real-time PCR data by the comparative C(T) method. Nat Protoc. 2008;3(6):1101-8. doi: 10.1038/nprot.2008.73. PMID 18546601
- [Background] Talbi S, Hamilton AE, Vo KC, Tulac S, Overgaard MT, Dosiou C, Le Shay N, Nezhat CN, Kempson R, Lessey BA, Nayak NR, Giudice LC. Molecular phenotyping of human endometrium distinguishes menstrual cycle phases and underlying biological processes in normo-ovulatory women. Endocrinology. 2006 Mar;147(3):1097-121. doi: 10.1210/en.2005-1076. Epub 2005 Nov 23. PMID 16306079
- [Background] Vitagliano A, Di Spiezio Sardo A, Saccone G, Valenti G, Sapia F, Kamath MS, Blaganje M, Andrisani A, Ambrosini G. Endometrial scratch injury for women with one or more previous failed embryo transfers: a systematic review and meta-analysis of randomized controlled trials. Fertil Steril. 2018 Sep;110(4):687-702.e2. doi: 10.1016/j.fertnstert.2018.04.040. PMID 30196966
- [Background] Yoo JY, Kim TH, Fazleabas AT, Palomino WA, Ahn SH, Tayade C, Schammel DP, Young SL, Jeong JW, Lessey BA. KRAS Activation and over-expression of SIRT1/BCL6 Contributes to the Pathogenesis of Endometriosis and Progesterone Resistance. Sci Rep. 2017 Jul 28;7(1):6765. doi: 10.1038/s41598-017-04577-w. PMID 28754906